CLINICAL TRIAL: NCT07158151
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Study Evaluating the Efficacy and Safety of RSS0393 Ointment in Adults With Mild to Moderate Atopic Dermatitis
Brief Title: A Phase II Trial of the Safety and Efficacy of RSS0309 Ointment in Adults With Atopic Dermatitis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Reistone Biopharma Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RSS0393Oint-202
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-08

CONDITIONS: Atopic Dermatitis of Adults

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group 1: RSS0393 ointment 0.05% (Experimental)
  Interventions: Drug: RSS0393 ointment
- Treatment group 2: RSS0393 ointment 0.01% (Experimental)
  Interventions: Drug: RSS0393 ointment
- Treatment group 3: RSS0393 ointment 0.03% (Experimental)
  Interventions: Drug: RSS0393 ointment
- Treatment group 4: RSS0393 ointment placebo (Sham Comparator)
  Interventions: Drug: RSS0393 ointment

INTERVENTIONS:
Drug: RSS0393 ointment — RSS0393 ointment 0.05%
  Arms: Treatment group 1: RSS0393 ointment 0.05%
Drug: RSS0393 ointment — RSS0393 ointment 0.01%
  Arms: Treatment group 2: RSS0393 ointment 0.01%
Drug: RSS0393 ointment — RSS0393 ointment 0.03%
  Arms: Treatment group 3: RSS0393 ointment 0.03%
Drug: RSS0393 ointment — RSS0393 ointment placebo
  Arms: Treatment group 4: RSS0393 ointment placebo

SUMMARY:
This study is ongoing to explore the efficacy and safety of different strengths of RSS0393 ointment in adults with atopic dermatitis

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old and ≤75 years old at screening.
2. History of atopic dermatitis ≥ 6 months.
3. BSA is between 3% and 20% (inclusive) and EASI score is ≥ 5 and vIGA-AD is 2 or 3.
4. The subjects signed informed consent before any study-related procedures began.

Exclusion Criteria:

1. Diagnosis of other dermatologic diseases at screening.
2. Subjects have other skin diseases or conditions that may affect the evaluation of the relevant endpoints of this study.
3. Subjects with any other persistent active autoimmune disease.
4. Subjects who have received topical medication for psoriasis within 14 days before baseline, or systemic medication or phototherapy for psoriasis within 28 days before baseline, or biological agents for psoriasis within a specified time before baseline.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2025-09-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with vIGA-AD success | Baseline, week 4
  The vIGA-AD is a static evaluation of qualitative overall AD severity. This global assessment scale is an ordinal scale with five severity grades (reported only in integers of 0 to 4 where 0 is clear). IGA sucess is defined as a vIGA-AD score of 'clear' or 'almost clear' plus at least 2-grade improvement from baseline

SECONDARY OUTCOMES:
Percentage of subjects with at least 75% reduction in the Eczema Area and Severity Index (EASI-75) | Up to 8 weeks
  EASI combines the assessment of the severity of lesions and the area affected into a single total score in the range 0 (no disease) to 72 (maximal disease).
Percentage of subjects with vIGA-AD of "clear" or "almost clear" | Up to 8 weeks
  The vIGA-AD is a static evaluation of qualitative overall AD severity. This global assessment scale is an ordinal scale with five severity grades (reported only in integers of 0 to 4 where 0 is clear).
The change of WI-NRS | Up to 8 weeks
  The Worst Itch Numerical Rating Scale (WI-NRS) will be determined by the subject's recording of daily assessment of worst itch over the past 24 hours.
Safety: treatment emergence adverse events | Up to 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided